CLINICAL TRIAL: NCT02452632
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Parallel-group, Placebo-Controlled Study to Assess the Efficacy and Safety of ASP1941 in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin and Sitagliptin
Brief Title: A Study to Assess the Efficacy and Safety of ASP1941 in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin and Sitagliptin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-2009
Record Dates: First submitted 2015-05-14; First posted 2015-05-22 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: ASP1941; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1941 group (Experimental): once daily over a 24 week treatment
  Interventions: Drug: ASP1941
- Placebo group (Placebo Comparator): once daily over a 24 week treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Other Names: ipragliflozin; Suglat
  Arms: ASP1941 group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ASP1941 50mg once daily in combination with metformin and sitagliptin against placebo in combination with metformin and sitagliptin over a 24 week treatment period in subjects with type 2 diabetes mellitus with inadequate glycemic control on metformin and sitagliptin.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with type 2 diabetes mellitus.
* Subject has an HbA1c value between 7.0% and 10.5 % at visit 1.
* Subject shows FPG (Fasting Plasma Glucose) value is less than 270mg/dL.
* Subject shows a BMI of 20.0 to 45.0 kg/m2.
* Subject is on stable diet and exercise program at least 8 weeks prior to study participation.
* Postmenopausal female or surgically sterile female or agree not to become pregnant.

Exclusion Criteria:

* Subject has type 1 diabetes mellitus.
* Subject has proliferative diabetic retinopathy.
* Subject has a history of clinically significant renal disease(s) such as renovascular occlusive disease, nephrectomy, or renal transplant.
* Subject has significant dysuria caused by a neurogenic bladder or a benign prostatic hypertrophy etc.
* Subject has a symptomatic urinary tract infection or genital infection.
* Subject has chronic disease(s) that require the continuous use of systemic corticosteroids or immunosuppressants.
* Subject has cardiovascular disease or cerebrovascular disease that may affect the administration of ASP1941 or its safety assessment in the opinion of the investigator or sub-investigator.
* Subject has uncontrollable psychiatric disorder(s) with medication.
* Male subject is not willing to use appropriate contraception during the study.
* Subject has severe infection, serious trauma, or perioperative subject.
* Subject has a malignant tumor or has a history of malignant tumor.
* Subject has severe gastrointestinal disease, or history of operation for serious gastrointestinal disease.
* Subject has diabetic ketoacidosis.
* Subject has lactic acidosis or has history of lactic acidosis.
* Subject has hepatitis or is a carrier of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or is positive for HIV-1 and/or HIV-2.
* Subject has a history of thyroid dysfunction and acute pancreatitis.
* Subject is on weight-loss program or weight-loss medication (e.g. orlistat, phentermine/topiramate, lorcaserin) within 12 weeks of study participation.
* Subject has a history of serious cardiac diseases (NYHA Class III to IV), congestive heart failure, arrhythmia in need of medical treatment.
* Subject has a history of cerebrovascular attack, unstable angina, myocardial infarction, angioplasty, within 52 weeks (364 days) of study participation.
* Subject has uncontrollable severe hypertension, i.e., systolic blood pressure of higher than 180 mmHg or diastolic blood pressure of higher than 110mmHg measured in a sitting position after a 5-minute rest.
* Subject has following AST or ALT value:

  * AST: Male > 100 U/L, Female > 80 U/L
  * ALT: Male > 102.5 U/L, Female > 82.5 U/L
* Subject has following serum creatinine value:

  * Creatinine: Male > 1.3 mg/dL, Female > 1.2 mg/dL
* Subject has estimated GFR values, of < 60 mL/min/1.73m2.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at the end of treatment | at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in Fasting plasma glucose at the end of treatment | at 24 weeks
Change from baseline in Fasting serum insulin at the end of treatment | at 24 weeks
Change from baseline in Body weight at the end of treatment | at 24 weeks
Change from baseline in Waist circumference at the end of treatment | at 24 weeks
Safety assessed by development of adverse events, vital signs, laboratory tests, and 12-lead ECG | up to 24 weeks
  ECG: Electrocardiogram
Number of subjects achieving the target HbA1c(<6.5% and <7.0%) at each visit | at 4, 8, 12, 16 and 24 weeks
Percentage of subjects achieving the target HbA1c(<6.5% and <7.0%) at each visit | at 4, 8, 12, 16 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Korea, Inc.
Locations (22):
- South Korea (22):
  - Site KR00019, Dong Gu Gwangju, Dong Gu Gwangju
  - Site KR00008, Gangwon-do, Gangwon-do
  - Site KR00020, Jeollabuk-do, Jeollabuk-do
  - Site KR00021, Kyungsangnam-do, Kyungsangnam-do
  - Site KR00002, Busan
  - Site KR00003, Busan
  - Site KR00007, Daegu
  - Site KR00011, Daegu
  - Site KR00018, Gyeonggi-do
  - Site KR00022, Gyeonggi-do
  - Site KR00014, Incheon
  - Site KR00001, Seoul
  - Site KR00004, Seoul
  - Site KR00005, Seoul
  - Site KR00006, Seoul
  - Site KR00009, Seoul
  - Site KR00010, Seoul
  - Site KR00012, Seoul
  - Site KR00013, Seoul
  - Site KR00016, Seoul
  - Site KR00017, Seoul
  - Site KR00015, Suwon

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=234